CLINICAL TRIAL: NCT00339443
Title: Calibration of Urine pH Strips for NCI Case-Control Studies on Bladder Cancer and Comparison of DNA Yields From Buccal Cells Collected Through Two Different Methods
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902040; 02-C-N040
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-19

CONDITIONS: Calibration
Keywords: Buccal Cells; Concordance; DNA Yields; pH Meter; Urine pH; Calibration

SUMMARY:
We propose to conduct a pilot study among 30 volunteers from the Division of Cancer Epidemiology and Genetics (DCEG) in order to: (1) select the urine pH strip that most closely correlates with urine pH measured by pH meter for the New England Bladder Cancer Study, (2) calibrate the urine pH strip that was used for the Spanish Bladder Cancer Study against pH measured by a pH meter, and (3) compare the DNA yields from buccal cells obtained from two different methods: mouthwash vs toothbrush-rinse method. Information collected from this pilot study will be used to select and optimize the sample collection protocols in the New England Bladder Cancer Study. At the time of enrollment, study participants will be asked to provide information on age, gender, height, weight, consumption of antacids and calcium supplements, and whether they ate, drank or brushed their teeth in the last hour previous to the buccal cells ample collection. In addition, they will have to measure their urine pH with four different pH strips twice a day (early morning and before dinner) for a week and record the measurements in a diary. During the same week, they will be asked to collect two spot urine samples each day from Monday to Thursday (early morning and before dinner), and one more on Friday morning, and bring them into work in a cooler. Also, they will be asked to collect a continuous 24-hour urine sample during one of the three first days of the week. Urine samples will e picked up by lab personnel from BioReliance, and pH will be measured at their laboratory with the four pH strips again and with a pH meter. Buccal cells sample collection will be completed during the first and the last day of the urine sample collection period. The first day, study participants will be asked to provide a water rinse sample after brushing the inside of their cheeks with a toothbrush, and a week later they will be asked to provide a mouth wash sample consisting of two consecutive rinses with Scope mouthwash. All samples and questionnaire data will be unlinked from personal identifiers after the sample collection is completed. Participants will be compensated with $100 for the inconvenience of participating in this complex study and for their time.

DETAILED DESCRIPTION:
We conducted a pilot study among 30 volunteers from the Division of Cancer Epidemiology and Genetics (DCEG) in order to: (1) select the urine pH strip that most closely correlates with urine pH measured by pH meter for the New England Bladder Cancer Study, (2) calibrate the urine pH strip that was used for the Spanish Bladder Cancer Study against pH measured by a pH meter, and (3) compare the DNA yields from buccal cells obtained from two different methods: mouthwash vs toothbrush-rinse method. At the time of enrollment, study participants were asked to provide information on age, gender, height, weight, consumption of antacids and calcium supplements, and whether they ate, drank or brushed their teeth in the last hour previous to the buccal cells sample collection. In addition, they measured their urine pH with four different pH strips twice a day (early morning and before dinner) for a week and record the measurements in a diary. During the same week, they were asked to collect two spot urine samples each day from Monday to Thursday (early morning and before dinner), and one more on Friday morning, and bring them into work in a cooler. Also, they were asked to collect a continuous 24-hour urine sample during one of the three first days of the week. Urine samples were picked up by lab personnel from BioReliance, and pH was measured at their laboratory with the four pH strips again and with a pH meter. Buccal cells sample collection was completed during the first and the last day of the urine sample collection period. The first day, study participants were asked to provide a water rinse sample after brushing the inside of their cheeks with a toothbrush, and a week later they were asked to provide a mouth wash sample consisting of two consecutive rinses with Scope mouthwash. All samples and questionnaire data was unlinked from personal identifiers after the sample collection was completed. Participants were compensated with $100 for the inconvenience of participating in this complex study and for their time. Information collected from this pilot study has been used to prepare manuscripts, as well as select and optimize the sample collection protocols in the New England Bladder Cancer Study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Members of the DCEG staff.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2001-11-06; Study Completion 2010-05-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States